CLINICAL TRIAL: NCT01196624
Title: Efficacy of Repetitive Transcranial Magnetic Stimulation Right Versus Left, With or Without Traumatic Stimuli in the Treatment of Posttraumatic Stress Disorder (PTSD) and Its Flashbacks
Brief Title: Repetitive Transcranial Magnetic Stimulation With Or Without Traumatic Stimuli in Post Traumatic Stress Disorder (PTSD)
Acronym: BSPTSDTMS2010
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beersheva Mental Health Center (Other Government)
Responsible Party: Principal Investigator, Joseph Levine, MD, psychiatrist, Beersheva Mental Health Center
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Diagnostic
Other Study IDs: BeershevaMHC - 4733CTIL
Record Dates: First submitted 2010-06-28; First posted 2010-09-08 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Flashbacks; Posttraumatic Stress Disorder
Keywords: PTSD; FLASHBACKS; TMS; EXPOSURE
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- TMS TO RT DLPF WITH EXPOSURE (Active Comparator): TMS TO RIGHT PREFRONTAL DORSOLATERAL BRAIN AREA WITH EXPOSURE
  Interventions: Device: rapid TMS, EXPOSURE TO TRAUMATIC STIMULI; Device: rapid TMS, EXPOSURE
- TMS TO RIGHT DLPF BRAIN AREA WITHOUT EXPOSURE (Active Comparator): TMS TO RIGHT DLPF BRAIN AREA WITHOUT EXPOSURE
  Interventions: Device: rapid TMS, EXPOSURE TO TRAUMATIC STIMULI; Device: rapid TMS, EXPOSURE
- TMS TO LEFT PREFRONTAL DORSOLATERAL BRAIN AREA WITH EXPOSURE (Active Comparator): TMS TO LEFT PREFRONTAL DORSOLATERAL BRAIN AREA WITH EXPOSURE
  Interventions: Device: rapid TMS, EXPOSURE TO TRAUMATIC STIMULI; Device: rapid TMS, EXPOSURE
- TMS TO LEFT DLPF BRAIN AREA WITHOUT EXPOSURE (Active Comparator): TMS TO LEFT DLPF BRAIN AREA WITHOUT EXPOSURE
  Interventions: Device: rapid TMS, EXPOSURE TO TRAUMATIC STIMULI; Device: rapid TMS, EXPOSURE

INTERVENTIONS:
Device: rapid TMS, EXPOSURE TO TRAUMATIC STIMULI — RAPID TMS, EXPOSURE TO TRAUMATIC STIMULI
Device: rapid TMS, EXPOSURE — apid TMS, EXPOSURE

SUMMARY:
Subjects

Forty consecutive patients fulfilling the DSM-IV diagnostic criteria for PTSD will be recruited from the inpatient and outpatient treatment programs at the Beer Sheva Mental Health Center. Patients will complet a course of 10 daily rTMS sessions.

After receiving a full explanation of the procedures, all subjects will sign a written informed consent statement approved by the Helsinki Ethics Committee of Ben-Gurion University.

Study Design

The study suggested here will recruit 40 patients with DSM-IV PTSD also demonstrating at least moderately severe flashbacks. Each of the subjects will be recruited randomly to one of 4 groups:

1. Right DLPF Rtms (10Hz) co-administered with neutral visual and/or auditori stimuli;
2. Right DLPF Rtms (10Hz) co-administered with visual and/or auditori traumatic stimuli mimicking experiences appearing during the patients flashbacks;
3. Left DLPF Rtms (10Hz) co-administered with neutral visual and or auditori stimuli;
4. Left DLPF Rtms (10Hz) co-administered with visual and/or auditori traumatic stimuli mimicking experiences appearing during the patients flashbacks;

Treatment Characteristics

rTMS will be performed with a Magstim stimulator (Magstim Company, Whitland, U.K.) The motor threshold was determined in each subject once, before treatment. This was defined as the lowest stimulation intensity capable of inducing a visible movement at least five times out of 10 stimulations.

The position of the right dorsolateral prefrontal cortex will be defined as 5 cm anterior (in a parasagittal line) to the motor cortex. The stimulus intensity will be 80% of the patient's motor threshold intensity.

Treatments will be given for 20 minutes per day over 10 working days. Both subjects received high-frequency rTMS) received 10 Hz for 2 seconds per train; the intertrain interval was 58 seconds. For each participant the stimulus was administered over the right dorsolateral prefrontal cortex.

Rating Scales

The ratings of PTSD symptoms, anxiety, and depression willm be carried out by an expert investigator who will be blind to the stimulation condition. The patients will be assessed at four time points-before TMS (baseline), at day 5, at day 10, and at day 24 (14 days after the intervention). The instruments used will be as follows:

The PTSD Checklist The Treatment Outcome PTSD Scale The Hamilton Anxiety Rating Scale The Hamilton Rating Scale for Depression PTSD symptoms were assessed by using the Hebrew version of the Clinician-Administered PTSD Scale.

DETAILED DESCRIPTION:
Subjects

Forty consecutive patients fulfilling the DSM-IV diagnostic criteria for PTSD (as assessed by the Structured Clinical Interview) will be recruited from the inpatient and outpatient treatment programs at the Beer Sheva Mental Health Center. Patients will complet a course of 10 daily rTMS sessions.

The exclusion criteria includ: substance use disorder, cardiac pacemaker implant, or a history of epilepsy, neurosurgery, or brain trauma. Patients suffering from chronic medical conditions of any sort will be excluded from the study.

After receiving a full explanation of the procedures, all subjects will sign a written informed consent statement approved by the Helsinki Ethics Committee of Ben-Gurion University.

Study Design

The study suggested here will recruit 40 patients with DSM-IV PTSD also demonstrating at least moderately severe flashbacks. Each of the subjects will be recruited randomly to one of 4 groups:

1. Right DLPF Rtms (10Hz) co-administered with neutral visual and/or auditori stimuli;
2. Right DLPF Rtms (10Hz) co-administered with visual and/or auditori traumatic stimuli mimicking experiences appearing during the patients flashbacks;
3. Left DLPF Rtms (10Hz) co-administered with neutral visual and or auditori stimuli;
4. Left DLPF Rtms (10Hz) co-administered with visual and/or auditori traumatic stimuli mimicking experiences appearing during the patients flashbacks;

Treatment Characteristics

rTMS will be performed with a Magstim stimulator (Magstim Company, Whitland, U.K.) having a circular coil with a 9-cm diameter.

The motor threshold will be determined in each subject once, before treatment. This will be defined as the lowest stimulation intensity capable of inducing a visible movement at least five times out of 10 stimulations.

The position of the right dorsolateral prefrontal cortex will be defined as 5 cm anterior (in a parasagittal line) to the motor cortex. The stimulus intensity will be 80% of the patient's motor threshold intensity.

Treatments will be given for 20 minutes per day over 10 working days subjects will receive high-frequency rTMS in a 10 Hz for 2 seconds per train; the intertrain interval will be 58 seconds. For each participant the stimulus will be administered over the right dorsolateral prefrontal cortex.

Rating Scales

The ratings of PTSD symptoms, anxiety, and depression willm be carried out by an expert investigator who will be blind to the stimulation condition. The patients will be assessed at four time points-before TMS (baseline), at day 5, at day 10, and at day 24 (14 days after the intervention). The instruments used will be as follows.

The PTSD Checklist is a 17-item self-report checklist of PTSD symptoms based closely on the DSM-IV criteria. The respondents rate each item from 1 ("not at all") to 5 ("extremely") to indicate the degree to which they have been bothered by that particular symptom over the past month. Thus, the total scores can range from 17 to 85.

The Treatment Outcome PTSD Scale is a clinician-rated instrument that measures the presence and severity of PTSD. This eight-item instrument measures symptoms that occur frequently within the PTSD population and is sensitive to the three major PTSD symptom dimensions (intrusive thoughts, avoidance behavior, and hyperarousal symptoms). Each symptom is rated on a defined step scale (0 to 4). Higher scores reflect greater severity on each measure.

The Hamilton Anxiety Rating Scale is a clinician-rated instrument that measures the presence and severity of anxiety. This instrument covers 14 symptoms. Each symptom is rated on a defined scale (0 to 4). Here, too, a higher numeric rating reflects greater symptom severity.

The Hamilton Rating Scale for Depression is a 23-item instrument that measures the presence and severity of depression. Each symptom is rated on a defined scale (0 to 4), whereby a higher numeric rating reflects greater symptom severity.

PTSD symptoms were assessed by using the Hebrew version of the Clinician-Administered PTSD Scale. This is a structured interview for assessing PTSD according to DSM-IV criteria. It quantifies symptom frequency and intensity for each of the criteria, yielding both a continuous measure of symptom severity and a dichotomous classification of PTSD status. A severity score for each symptom is calculated by summing the frequency and intensity scores. Thus, the total range of the instrument is 0-136. If a particular symptom was not present, the individual item was automatically scored as zero, as a default option. The Hebrew version of the scale has been extensively used and validated

The questionnaires will be filled out in the presence of an interviewer, and the subjects will be assisted in answering the questions if necessary. The interviewer will made sure that all subjects clearly understood the content of each item and the different aspects of the various component questions.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients fulfilling the DSM-IV diagnostic criteria for PTSD (as assessed by the Structured Clinical Interview) will be recruited from the inpatient and outpatient treatment programs at the Beer Sheva Mental Health Center.

Exclusion Criteria:

Subjects

The exclusion criteria includ:

* substance use disorder, cardiac pacemaker implant, or a history of epilepsy, neurosurgery, or brain trauma.
* Patients suffering from chronic medical conditions of any sort will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
flashback severity, CAPS score | the study will be held for 1-2 years

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Levine, Associate Professor, Principal Investigator — Beersheva mental Health Center, Israel; Nimrod Grisaru, Principal Investigator — Beersheva Mental Health Center
Locations (1):
- Beersheva mental Health Center, Beersheva,, Israel